CLINICAL TRIAL: NCT05042375
Title: A Randomized, Open-Label, Controlled, Multi-center Phase Ⅲ Study of Camrelizumab Combined With Famitinib Malate Versus Pembrolizumab in Treatment Naïve Subjects With PD-L1-Positive Recurrent or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Trial of Camrelizumab Combined With Famitinib Malate in Treatment Naïve Subjects With PD-L1-Positive Recurrent or Metastatic Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-III-331
Record Dates: First submitted 2021-09-01; First posted 2021-09-13 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-10

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — camrelizumab; famitinib; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Camrelizumab Combined with Famitinib Malate versus Pembrolizumab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- camrelizumab + famitinib (Experimental)
  Interventions: Drug: camrelizumab + famitinib
- pembrolizumab (Experimental)
  Interventions: Drug: pembrolizumab
- camrelizumab (Experimental)
  Interventions: Drug: camrelizumab

INTERVENTIONS:
Drug: camrelizumab + famitinib — Camrelizumab for injection, 200 mg; Famitinib malate capsules, 20 mg.
  Arms: camrelizumab + famitinib
Drug: pembrolizumab — pembrolizumab 200 mg.
  Arms: pembrolizumab
Drug: camrelizumab — Camrelizumab for injection, 200 mg.
  Arms: camrelizumab

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of camrelizumab combined with famitinib malate vs. pembrolizumab in treatment naïve subjects with programmed death-ligand 1(PD-L1)-positive recurrent or metastatic non-small cell lung cancer (NSCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Have a histologically or cytologically confirmed diagnosis of metastatic NSCLC (stage IV according to the TNM staging criteria [8th edition] published by the International Association for the Study of Lung Cancer [IASLC]), or NSCLC that recurs after curable surgery, radiotherapy, or radiochemotherapy.
2. Have measurable disease based on RECIST v1.1.
3. ECOG PS score: 0-1.
4. Have a life expectancy of at least 3 months.
5. Non-surgically sterilized female subjects or women of childbearing potential must be negative for a serum pregnancy test within 3 days prior to the first dose and must be non-lactating. Female subjects of childbearing potential and male subjects with partners of childbearing potential must agree to take highly effective contraceptive measures during the study period and within 6 months after the last dose of study drugs.
6. Have voluntarily agreed to participate by giving written informed consent for the study, have good compliance, and cooperate with follow-up visits.

Exclusion Criteria:

1. Accompanied with EGFR activating mutation, ALK fusion gene positive or ROS1 mutation.
2. Have uncontrolled clinically symptomatic pleural effusion, pericardial effusion, or ascites.
3. Have known history of prior malignancy in the past 3 years.
4. Have had an allogeneic tissue/solid organ transplant.
5. Have active pulmonary tuberculosis.
6. Have clinical symptoms of the heart or heart diseases that are not well controlled.
7. Have hypertension which cannot be well controlled by antihypertensives
8. Urinalysis has indicated that the urine protein is ≥ ++ and quantitative test of urine protein has confirmed that the 24-h urine protein is > 1.0 g.
9. Have a thrombosis tendency or are currently receiving thrombolysis/anticoagulation therapy.
10. Have received major surgery within 4 weeks prior to randomization; or palliative radiotherapy within 2 weeks prior to randomization; or have not recovered from the toxicities and/or complications of previous interventions to NCI-CTCAE Grade ≤ 1.
11. Have known history of arterial/venous thrombosis within 6 months prior to randomization, such as cerebrovascular accidents, deep vein thrombosis and pulmonary embolism.
12. Have received prior therapy with anti-PD-1/PD-L1 monoclonal antibodies, anti-CTLA-4 monoclonal antibodies, or small molecule VEGFR inhibitors.
13. Have known allergies to other monoclonal antibodies or any component of famitinib.
14. Are currently participating and receiving study therapy or have participated in a study and received the last dose of study drug within 4 weeks (or 5 half-lives of the study drug) prior to randomization.
15. Have other potential factors that may affect the study results or result in the premature discontinuation as determined by the investigator, such as alcoholism, drug abuse, substance abuse, other serious diseases (including mental illness) requiring concomitant treatment, serious laboratory abnormalities, or family or social factors that could affect the safety of medication.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS assessed by BIRC | up to 3 years
  Progression-Free-Survival, defined as the time from randomization to the first occurrence of disease progression as determined by IRC with use of RECIST v1.1 or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
PFS assessed by investigator | up to 3 years
  Progression-Free-Survival
ORR | up to 3 years
  Objective Response Rate, determined using RECIST v1.1 criteria, defined as best overall response (CR or PR) across all assessment time points
DCR | up to 3 years
  Disease Control Rate, determined using RECIST v1.1 criteria
DoR | up to 3 years
  Duration of Response, determined using RECIST v1.1 criteria
TTF | up to 3 years
  Time to Treatment Failure, defined as the time from randomization to treatment discontinuation.
AEs+SAEs | from the first drug administration to within 90 days for the last SHR-1210 dose
  Adverse Events and Serious Adverse Events
OS | up to 4 years
  OS is the time interval from the date of randomization to death due to any reason or lost of follow-up

CONTACTS AND LOCATIONS:
Locations (80):
- China (80):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Chest Hospital, Hefei, Anhui
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital Of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - ChongQing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The Second Affiliated Hospital of Xiamen Medical College, Xiamen, Fujian
  - The People's Hospital of Gaozhou, Gaozhou, Guangdong
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Meizhou People's Hospital (Huangtang Hospital), Meizhou, Guangdong
  - Shantou Central Hospital, Shantou, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Hainan General Hospital, Haikou, Hainan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - North China University Of Science And Technology Affiliated Hospital, Tangshan, Hebei
  - Xingtai People's Hospital, Xingtai, Hebei
  - Haerbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang Cancer Hospital, Anyang, Henan
  - The First Affiliated Hosptial of Henan University of Science & Technology, Luoyang, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Shiyan Taihe Hospital, Shiyan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Army Medical Center of PLA, Changsha, Hunan
  - Hunan Cancer Hospital-Thoracic Medicine Department I, Changsha, Hunan
  - Hunan Cancer Hospital-Thoracic Medicine Department Ⅱ, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - Shaoyang Central Hospital, Shaoyang, Hunan
  - Zhuzhou Central Hospital, Zhuzhou, Hunan
  - Affiliated Drum Tower Hospital, Medical School of Nanjing University, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Affiliated Hospital of JiangNan University, Wuxi, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Chifeng City Hospital, Chifeng, Neimenggu
  - The Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Neimenggu
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Cancer Hospital&Institute, Jinan, Shandong
  - The Affiliated of Qingdao University, Qingdao, Shandong
  - LinYi Cancer Hospital, Linyi, Shangdong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Baoji Central Hospital, Baoji, Shanxi
  - Changzhi People's Hospital, Changzhi, Shanxi
  - General Hospital of TISCO, Taiyuan, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - The Second Affiliated Hospital of Air Force Military University Tangdu Hospital, Xi’an, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Yibin Second People's Hospital, Yibin, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Hangzhou Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital, College of Medicine, Zhejiang University of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - ZheJiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided